CLINICAL TRIAL: NCT02434952
Title: The Tolerability and Safety of Low Dose Primaquine for Transmission Blocking in Symptomatic Falciparum Infected Cambodians
Brief Title: Safety and Tolerability of Low Dose Primaquine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Malaria Consortium (Other)
Collaborators: National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other); Institute Pasteur, Cambodia (Unknown); World Health Organization (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 015NECHR
Record Dates: First submitted 2014-09-11; First posted 2015-05-06 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Malaria, Falciparum; G6PD Deficiency
Keywords: Malaria, Falciparum; G6PD deficiency; Primaquine; Asia
MeSH Terms: conditions — Malaria, Falciparum; Glucosephosphate Dehydrogenase Deficiency | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DHA PP plus primaquine, G6PD deficiency (Experimental): Standard Dihydroartemisinin piperaquine (DHA PP) dosing according to national guidelines, oral administration of one dose per day for three consecutive days. Target dosing is 2-4 mg/kg for DHA and 20 mg/kg for PP. Children (<30kg) will receive tablets of 20mg DHA and 160mg PP, while adults will receive tablets of 40mg DHA and 320mg PP.
  Target dose of 0.25mg/kg primaquine given orally with first dose only of DHA PP, dosing by weight for children <18 years and standard 15mg primaquine dose for all adults ≥18 years. Small children (<25kg) will receive a primaquine suspension, adults receive 7.5mg or 15mg primaquine tablets.
  Interventions: Drug: Dihydroartemisinin piperaquine (DHA PP); Drug: Primaquine
- DHA PP plus primaquine, G6PD normal (Active Comparator): Standard Dihydroartemisinin piperaquine (DHA PP) dosing according to national guidelines, oral administration of one dose per day for three consecutive days. Target dosing is 2-4 mg/kg for DHA and 20 mg/kg for PP. Children (<30kg) will receive tablets of 20mg DHA and 160mg PP, while adults will receive tablets of 40mg DHA and 320mg PP.
  Target dose of 0.25mg/kg primaquine given orally with first dose only of DHA PP, dosing by weight for children <18 years and standard 15mg primaquine dose for all adults ≥18 years. Small children (<25kg) will receive a primaquine suspension, adults receive 7.5mg or 15mg primaquine tablets.
  Interventions: Drug: Dihydroartemisinin piperaquine (DHA PP); Drug: Primaquine
- DHA PP alone, G6PD deficiency (Active Comparator): Standard Dihydroartemisinin piperaquine (DHA PP) dosing according to national guidelines, oral administration of one dose per day for three consecutive days. Target dosing is 2-4 mg/kg for DHA and 20 mg/kg for PP. Children (<30kg) will receive tablets of 20mg DHA and 160mg PP, while adults will receive tablets of 40mg DHA and 320mg PP.
  Interventions: Drug: Dihydroartemisinin piperaquine (DHA PP)
- DHA PP alone, G6PD normal (Active Comparator): Standard Dihydroartemisinin piperaquine (DHA PP) dosing according to national guidelines, oral administration of one dose per day for three consecutive days. Target dosing is 2-4 mg/kg for DHA and 20 mg/kg for PP. Children (<30kg) will receive tablets of 20mg DHA and 160mg PP, while adults will receive tablets of 40mg DHA and 320mg PP.
  Interventions: Drug: Dihydroartemisinin piperaquine (DHA PP)

INTERVENTIONS:
Drug: Dihydroartemisinin piperaquine (DHA PP)
  Other Names: Duo-Cotecxin; Eurartesim
Drug: Primaquine
  Arms: DHA PP plus primaquine, G6PD deficiency; DHA PP plus primaquine, G6PD normal

SUMMARY:
In Cambodia, falciparum is becoming more difficult to treat because drugs are becoming less effective. The investigators can help to try to prevent the spread of this resistant malaria by adding a drug that will make it more difficult for the mosquito to drink up the malaria in people's blood. If the mosquito cannot drink up the malaria, then the malaria cannot develop in the mosquito so it will not be able to inject malaria back into people when it bites. The drug the investigators will use is called primaquine.

Primaquine commonly causes the red cells in the blood to break apart if they are weak. Red cells need enzymes to work properly and weak red cells have low amounts of an enzyme called glucose 6 phosphate dehydrogenase (G6PD). The investigators want to know if treating malaria with primaquine will be safe for the red cells. To do this study, the investigators need to know if a subject has low G6PD or not.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 year
* Presentation with a confirmed fever (≥ 38⁰C axilla or ≥ 37.5⁰C aural) or history of fever in previous 48 hours +/- other clinical features of uncomplicated malaria
* Plasmodium falciparum monoinfection ≥ 1 asexual form / 500 white blood cells
* Informed consent (written/verbal) provided by patient or relative/legal guardian
* Signed Assent form for children aged 12 to < 18 years

Exclusion Criteria:

* Clinical signs of severe malaria or danger signs
* Pregnant or breast feeding
* Unable or unwilling to take a pregnancy test (for women of child-bearing age)
* Women intending to become pregnant in the next 3 months
* Allergic to primaquine or DHA PP
* Patients taking drugs known to cause acute intravascular haemolytic anaemia (AIHA) in G6PD deficiency e.g. dapsone, nalidixic acid
* Patients on treatment for a significant illness e.g. HIV, tuberculosis (TB) treatment, steroids
* On drugs that could interfere with anti-malarial pharmacokinetics like antiretrovirals, cimetidine, ketoconazole, antiepileptic drugs, rifampicin

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Haemoglobin concentration | Day 7
  Compare haemoglobin concentrations in g/dL between the G6PD deficient arm given DHA PP plus primaquine, and the G6PD normal arm receiving the same regimen

SECONDARY OUTCOMES:
Determine G6PD enzyme activity | Day 0
  Quantitative G6PD testing among all participants using the G6PD enzyme assay from Trinity Biologicals, USA, yielding G6PD enzyme results in U/g Hb.
Assess usefulness of field adapted WHO haemoglobin colour card vs. Hemocue | Day 0
  Comparison of quantitative (HemoCue, g/dL HB) and qualitative (WHO haemolglobin colour card) estimates of haemoglobin concentration
Assess usefulness of rapid test for G6PDd in predicting acute intravascular haemolysis | Day 0
  Comparison of rapid G6PD test (AccessBio, USA) qualitative result against quantitative G6PD assay to determine predictive value for clinically significant haemolysis
Proportion patients with ≥25% change in haemoglobin as a marker of intravascular haemolysis | Change from Day 0 to Day 7
  Comparing across all 4 arms: proportion of all patients with fractional change in haemoglobin ≥25% from day 0 to day 7
Plasma haemoglobin concentration as a marker of intravascular haemolysis | Day 7
  Comparing across all 4 arms: plasma haemoglobin concentration at day 7
Urine colour change as a marker of intravascular haemolysis | Change from Day 0 to Day 7
  Change in urine colour grade from day 0 to day 7 (Hillmen, Hall et al. 2004)
Fractional change in haemoglobin as a marker of intravascular haemolysis | Change from Day 0 to Day 7
  Comparing across all 4 arms: fractional change in haemoglobin on day 7 vs. day 0
Clearance rate of primaquine | Day 0-7
  Primaquine elimination clearance rate, modelled from population pharmacokinetic data from all patients receiving at least one dose of DHA PP + PQ
Half life of primaquine | Day 0-7
  Primaquine terminal elimination half life, modelled from population pharmacokinetic data from all patients receiving at least one dose of DHA PP + PQ
Primaquine volume of distribution | Day 0-7
  Primaquine apparent volume of distribution (Vd), modelled from population pharmacokinetic data from all patients receiving at least one dose of DHA PP + PQ
Clearance rate of piperaquine | Day 0-28
  Piperaquine elimination clearance rate, modelled from population pharmacokinetic data from all patients receiving at least one dose of DHA PP +/- PQ
Half life of piperaquine | Day 0-28
  Piperaquine terminal elimination half life, modelled from population pharmacokinetic data from all patients receiving at least one dose of DHA PP +/- PQ
Piperaquine volume of distribution | Day 0-28
  Piperaquine apparent volume of distribution (Vd), modelled from population pharmacokinetic data from all patients receiving at least one dose of DHA PP +/- PQ
Peak plasma concentration (Cmax) of primaquine | Day 0-7
  Cmax taken directly from population pharmacokinetic data from all patients receiving at least one dose of DHA PP + PQ
Peak plasma concentration (Cmax) of piperaquine | Day 0-28
  Cmax taken directly from population pharmacokinetic data from all patients receiving at least one dose of DHA PP +/- PQ
Time to primquine peak plasma concentration (Tmax) | Day 0-7
  Tmax taken directly from population pharmacokinetic data from all patients receiving at least one dose of DHA PP + PQ
Time to piperaquine peak plasma concentration (Tmax) | Day 0-28
  Tmax taken directly from population pharmacokinetic data from all patients receiving at least one dose of DHA PP +/- PQ
Area under the plasma concentration versus time curve - primaquine | Day 0-7
  Modelled from population pharmacokinetic data from all patients receiving at least one dose of DHA PP + PQ
Area under the plasma concentration versus time curve - piperaquine | Day 0-28
  Modelled from population pharmacokinetic data from all patients receiving at least one dose of DHA PP +/- PQ

CONTACTS AND LOCATIONS:
Overall Officials: Dysoley Lek, MD, Principal Investigator — National Centre for Parasitology, Entomology and Malaria Control, Cambodia
Locations (1):
- Ratanakiri Provincial Hospital, Ratanakiri, Ratanakiri, Cambodia

REFERENCES:
- [Derived] Vantaux A, Kim S, Piv E, Chy S, Berne L, Khim N, Lek D, Siv S, Mukaka M, Taylor WR, Menard D. Significant Efficacy of a Single Low Dose of Primaquine Compared to Stand-Alone Artemisinin Combination Therapy in Reducing Gametocyte Carriage in Cambodian Patients with Uncomplicated Multidrug-Resistant Plasmodium falciparum Malaria. Antimicrob Agents Chemother. 2020 May 21;64(6):e02108-19. doi: 10.1128/AAC.02108-19. Print 2020 May 21. PMID 32179526
- [Derived] Dysoley L, Kim S, Lopes S, Khim N, Bjorges S, Top S, Huch C, Rekol H, Westercamp N, Fukuda MM, Hwang J, Roca-Feltrer A, Mukaka M, Menard D, Taylor WR. The tolerability of single low dose primaquine in glucose-6-phosphate deficient and normal falciparum-infected Cambodians. BMC Infect Dis. 2019 Mar 12;19(1):250. doi: 10.1186/s12879-019-3862-1. PMID 30871496
- See also: Malaria Consortium — http://www.malariaconsortium.org/
- See also: National Centre for Parasitology, Entomology and Malaria Control Program, Cambodia — http://www.cnm.gov.kh/